CLINICAL TRIAL: NCT02453932
Title: A Phase III, Multicenter, Randomized, Double-blind, Positive /Placebo Controlled, Parallel, Three Arms Study of Tianzhi Granule in Mild to Moderate Vascular Dementia
Brief Title: Efficacy and Safety of Tianzhi Granule in Mild to Moderate Vascular Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, MD，PhD, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012ZX09104-203
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Vascular Dementia
Keywords: Vascular dementia; Tianzhi granule; Herbal medicine; Randomized controlled trial; Three arms
MeSH Terms: conditions — Dementia, Vascular | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tianzhi granule (Experimental): Tianzhi granule and placebo identified to donepezil
  Interventions: Drug: Tianzhi granule and placebo identified to donepezil
- Donepezil (Active Comparator): Donepezil and placebo identified to Tianzhi granule
  Interventions: Drug: Donepezil and placebo identified to Tianzhi granule
- Placebo (Placebo Comparator): Placebo identified toTianzhi granule and placebo identified to donepezil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tianzhi granule and placebo identified to donepezil — 1 pack Tianzhi granule (5g), 3 times per day and placebo identified to donepezil, 1 pill per day for 24 weeks
  Arms: Tianzhi granule
Drug: Donepezil and placebo identified to Tianzhi granule — donepezil 5mg per day and placebo identified to Tianzhi granule (5g, 3 times per day) for 24 weeks
  Arms: Donepezil
Drug: Placebo — placebo identified to Tianzhi granule (5g, 3 times per day) and placebo identified to donepezil ,1 pills per day for 24 weeks
  Arms: Placebo

SUMMARY:
This ongoing study aimed to evaluate the efficacy and safety of Tianzhi granule in mild to moderate vascular dementia in a more reasonable design.

DETAILED DESCRIPTION:
This study is a 24-weeks, multicenter, randomized, double-blind, double- placebo, parallel controlled phase III trial being carried out in 23 centers around China. The study population includes mild to moderate VaD patients (planned a total of 630) aged 45-85 in both gender. Participants will be randomly allocated to TZK (15g/d) and placebo identified to donepezil, donepezil (5mg/d) and placebo identified to TZK, or placebo identified to TZK and placebo identified to donepezil for a 24-weeks double-blind treatment period . The primary outcome measure is change from baseline in the Vascular Dementia Assessment Scale-Cognitive Subscale and Clinician's Interview-Based Impression of Change-Plus carer Interview. The secondary outcomes are changes from baseline in the Mini-Mental State Examination, Activity of Daily Living Scale, Clock Drawing Test, Trail Making Test and Neuropsychiatric Inventory. Safety is being assessed by observing side effects and adverse reaction during the entire treatment period. Statistical analysis will be conducted according to per-protocol population and intend-to-treat population and the safety will be analyzed in safety set.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients meeting the diagnostic criteria probable VaD established according to the Diagnostic and Statistical Manual of Mental Disorders (fourth edition) （DSM-Ⅳ） and the National Institute of Neurological Disorders and Stroke and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS-AIREN)were eligible to participate,
* diagnosis of mild to moderate vascular dementia;
* Chinese-speaking patients aged ≥45 and≤85 years old in both gender;
* weighing between 45 and 90kg;
* fully conscious;
* MMSE score of≤26 and ≥14;
* HIS score of ≥7;
* adequate vision and hearing ability to complete all study tests;
* with a stable caregiver.

Exclusion Criteria:

Patients will be excluded from the enrollment if they meet any of the followings:

* a medical history of other dementia types, like Alzheimer's disease, Parkinson's disease dementia, Huntington disease, Normal pressure hydrocephalus, et al;
* major depression (HAMD for 17 items>17) or psychotic disorder;
* acute stage of cerebral hemorrhage or subarachnoid hemorrhage;
* hypothyroidism;
* drug or alcohol abuse;
* epilepsy history; myasthenia gravis history;
* severe cardiovascular disease(severe arrhythmia with heart rate≥100 or≤60 times per min, left bundle branch block, myocardial infarction within 3 months, systolic pressure≥180mmHg or ≤90mmHg);
* severe liver or kidney dysfunction (alanine aminotransferase>60 IU/L, aspartate transaminase>60 IU/L or serum creatinine >266μmol/L);
* severe asthma or chronic obstructive pulmonary disease;
* gastrointestinal tract obstruction or severe peptic ulcer; glaucoma;
* administration of cholinesterase inhibitors, memantine or nimodipine in the last month;
* use of sympathomimetic agent, antihistamine drug, antianxiety drugs or tranquilizer within 48h before assessment;
* use of antipsychotic drugs within 72h before assessment;
* participation in other clinical trials; allergic history to any type of medication used in this study.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2013-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes of Vascular Dementia Assessment Scale-Cognitive Subscale(VADAS-cog) from baseline after 24 weeks' intervention | week 0, 4, 12, 24
  Cognition : VaDAS-cog is a revision of the ADAS-cog to be a better measure in vascular conditions. The original ADAS-cog developed by Rosen et al., measures cognitive performance by combining ratings of 11 items. The cognitive domains mainly addressed by ADAS-cog are memory (short term), language, ability to orientate (reflects memory), construction/planning of simple designs and performance. In addition to ADAS-cog, the VaDAS-cog comprises additional frontal lobe tests reflecting attention, working memory, executive function, and verbal fluency.The VADAS-cog will conducted at baseline, 4weeks, 12weeks, 24weeks
Changes of Clinician's Interview-Based Impression of Change-Plus carer Interview(CIBIC-plus) from baseline after 24 weeks' intervention | week 0, 4, 12, 24
  Overall clinical response: CIBIC-plus is a 7-point scale which provides an index of clinically important change for dementia patients. It is a global measure of detectable change in concentration, orientation, memory, language, behavior, initiative and activities of daily living, usually requiring separate interviews with patients and caregivers,the CIBIC-plus will be conducted at baseline, 4weeks, 12weeks, 24weeks

SECONDARY OUTCOMES:
Changes of Mini-Mental State Examination(MMSE) from baseline after 24 weeks' treatment | week 0, 4, 12, 24
  Global cognition will be assessed by the MMSE,which will be conducted at baseline, 4weeks, 12weeks, 24weeks.
Changes of Activity of Daily Living Scale(ADL) from baseline after 24 week's intervention | week 0, 4, 12, 24
  Function:The ADL mainly used to measure the basic activities of daily living (or self-care) and the instrumental activities of daily living. The ADL scale can be divided to Physical Self-Maintenance Scale (PSMS) and the instrumental activities of daily living (IADL). The PSMS relate to physical activities, such as toileting, mobility, dressing and bathing , and the IADL contains 8 items ,such as shopping, cooking, doing laundry, handling finances, using telephone, mode of transportation, responsibility for own medication and housekeeping.The ADL wil be conducted baseline, 4weeks, 12weeks, 24weeks
Changes of Clock Drawing Test(CDT) from baseline after 24 week's intervention | week 0, 4, 12, 24
  Executive function and Visuospatial function : the CDT scale will be conducted at baseline, 4weeks, 12weeks, 24weeks.
Changes of Trail Making Test (TMT) from baseline after 24 week's intervention | week 0, 4, 12, 24
  Executive function: The TMT scale will be conducted at baseline, 4weeks, 12weeks, 24weeks.
Changes of Neuropsychiatric Inventory(NPI) from baseline after 24 weeks' intervention | week 0, 4, 12, 24
  Changes in psychological symptom: NPI is used throughout the study to assess changes in psychological symptom,the NPI will be conducted at baseline, 4 weeks, 12 weeks, 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Tian, MD,PhD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shi J, Wei M, Ni J, Sun F, Sun L, Wang J, Yu T, Wang K, Lv P, Wang Y, Zhang Y, Gao X, Gao X, Luo B, Mao S, Zhang B, Ren X, Yu F, Hu W, Yin P, Wu N, Liu X, Bi Q, Wang Y, Tian J; CHASE Study Group. Tianzhi granule improves cognition and BPSD of vascular dementia: a randomized controlled trial. J Transl Med. 2020 Feb 13;18(1):76. doi: 10.1186/s12967-020-02232-z. PMID 32054507